CLINICAL TRIAL: NCT04108195
Title: A Phase 1b Study of Subcutaneous Daratumumab Regimens in Combination With Bispecific T Cell Redirection Antibodies for the Treatment of Subjects With Multiple Myeloma
Brief Title: A Study of Subcutaneous Daratumumab Regimens in Combination With Bispecific T Cell Redirection Antibodies for the Treatment of Participants With Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108620; 64407564MMY1002 (Other: Janssen Research & Development, LLC); 2019-000330-19 (EudraCT Number); 2023-503468-17-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; talquetamab; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will be assigned to either a combination of 1) daratumumab plus teclistamab or 2) daratumumab plus talquetamab or 3) daratumumab plus talquetamab plus pomalidomide or 4) daratumumab plus teclistamab plus pomalidomide.
  Interventions: Drug: Daratumumab; Drug: Talquetamab; Drug: Teclistamab; Drug: Pomalidomide
- Part 2: Dose Expansion (Experimental): Participants will be treated with the RP2D(s) for selected treatment combinations determined in Part 1.
  Interventions: Drug: Daratumumab; Drug: Talquetamab; Drug: Teclistamab; Drug: Pomalidomide

INTERVENTIONS:
Drug: Daratumumab — Participants will receive daratumumab.
  Other Names: JNJ-54767414, Darzalex
Drug: Talquetamab — Participants will receive talquetamab.
  Other Names: JNJ-64407564
Drug: Teclistamab — Participants will receive teclistamab.
  Other Names: JNJ-64007957
Drug: Pomalidomide — Participants will receive pomalidomide.

SUMMARY:
The purpose of this study is to identify recommended Phase 2 doses (RP2Ds) for each treatment combination (between daratumumab plus talquetamab and teclistamab plus daratumumab with or without pomalidomide) and to characterize the safety of each RP2D for selected treatment combinations.

DETAILED DESCRIPTION:
Multiple myeloma is a malignant plasma cell disorder characterized by osteolytic lesions, increased susceptibility to infections, hypercalcemia, and renal failure. Overall rationale of study is that daratumumab in combination with talquetamab or teclistamab with or without pomalidomide may lead to enhanced clinical responses in treatment of relapsed or refractory multiple myeloma through multiple mechanisms of action. Daratumumab is human immunoglobulin G1 kappa monoclonal antibody (IgG1k) that binds with high affinity to a unique epitope on cluster of differentiation 38 (CD38) in a variety of hematological malignancies including multiple myeloma. Talquetamab and teclistamab are bispecific T cell redirection antibodies. Talquetamab binds to cluster of differentiation 3 (CD3) receptor complex on T cells and to G protein-coupled receptor family C group 5-member D (GPRC5D), a 7-transmembrane receptor protein on plasma cells and teclistamab binds to human and cynomolgus-CD3 and B cell maturation antigen (BCMA). Purpose of study is to evaluate safety of daratumumab in combination with talquetamab and teclistamab with or without pomalidomide, and to evaluate preliminary antitumor activity of each combination. Study consists of a screening period, treatment period (Part 1: dose escalation and Part 2: dose expansion), a Post-treatment Follow-up Period (after the last dose of study drug and will continue for up to 16 weeks for each subject), and a Long-term Extension Period. The study will end when one of the following occurs: 1) the study drug has received marketing authorization and, if regionally applicable, government reimbursement is available; 2) a long-term extension rollover study has commenced for participants who are still benefiting from study treatment as determined by their investigator; or 3) all participants have discontinued study treatment. Total duration of study is approximately 5 years and 6 months. Efficacy, safety, pharmacokinetics (PK), immunogenicity, and biomarkers will be assessed at specified time points. Participants safety will be monitored throughout study by Study Evaluation Team (SET). SET consists of members of sponsor's study team and participating investigators.

ELIGIBILITY:
Inclusion Criteria:

* Documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Must have either of the following: a) received at least 3 prior lines of therapy including a proteasome inhibitor (PI) (greater than or equal to [>=] 2 cycles or 2 months of treatment) and an immunomodulatory drug (IMiD) (>=2 cycles or 2 months of treatment) in any order during the treatment or b) disease that is double refractory to a PI and an IMiD
* Measurable disease at screening as defined by any of the following: Serum monoclonal protein (M-protein) level >=1.0 grams per deciliter (g/dL) (in non- immunoglobulin G (IgG) myeloma, an M-protein level >=0.5 g/dL); or Urine M-protein level >=200 milligrams (mg)/24 hours; or Light chain multiple myeloma: Serum immunoglobulin (Ig) free light chain (FLC) >=10 milligrams per deciliter (mg/dL) and abnormal serum Ig kappa lambda FLC ratio
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1 at screening and at Cycle 1, Day 1 predose
* Female participants of childbearing potential must have a negative highly-sensitive serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test (less than [<] 5 international units per milliliter [IU/mL]) at screening and a negative urine or serum pregnancy test within 1 day before the first dose of study drug

Exclusion Criteria:

* Treatment in the prior 3 months with an anti- cluster of differentiation 38 (CD38) therapy (example, daratumumab), or discontinuation of a prior anti-CD38 therapy at any time due to an adverse event related to the anti-CD38 therapy
* Live, attenuated vaccine within 4 weeks prior to the first dose of study drug unless approved by sponsor
* Active Central nervous system involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, brain magnetic resonance imaging (MRI) and lumbar cytology are required
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded
* Active hepatitis C infection as measured by positive hepatitis C virus- ribonucleotide (HCV)-RNA testing. Participants with a history of Hepatitis C virus antibody positivity must undergo HCV-RNA testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Dose Limiting Toxicity (DLT) | Up to 52 Weeks
  The dose limiting toxicities are based on drug related adverse events and defined as any of the following events: hematological or non-hematological toxicity of grade 3 or higher.
Part 1: Number of Participants With Dose Limiting Toxicity by Severity | Up to 52 Weeks
  The dose limiting toxicities are based on drug related adverse events and defined as any of the following events: hematological or non-hematological toxicity of grade 3 or higher.
Part 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 48 Weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, and suspects transmission of any infectious agent via a medicinal product.
Part 2: Number of Participants With Adverse Events and SAEs by Severity | Up to 48 Weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, and suspects transmission of any infectious agent via a medicinal product.

SECONDARY OUTCOMES:
Serum Concentration of Daratumumab | Up to 52 Weeks
  Serum concentration of daratumumab will be assessed.
Serum Concentration of Talquetamab | Up to 52 Weeks
  Serum concentration of talquetamab will be assessed.
Serum Concentration of Teclistamab | Up to 52 Weeks
  Serum concentration of teclistamab will be assessed.
Biomarker Assessment of Daratumumab | Up to Cycle 7 Day 1 (each cycle of 28-days)
  Serum cytokine concentrations will be measured at the time of drug infusion of daratumumab for biomarker assessment.
Biomarker Assessment of Talquetamab | Up to Cycle 7 Day 1 (each cycle of 28-days)
  Serum cytokine concentrations will be measured at the time of drug infusion of talquetamab for biomarker assessment.
Biomarker Assessment of Teclistamab | Up to Cycle 7 Day 1 (each cycle of 28-days)
  Serum cytokine concentrations will be measured at the time of drug infusion of teclistamab for biomarker assessment.
Number of Participants With Anti-Drug Antibodies to Daratumumab | Up to 52 Weeks
  Number of participants with anti-drug antibodies to daratumumab will be assessed.
Number of Participants With Anti-Drug Antibodies to Talquetamab | Up to 52 Weeks
  Number of participants with anti-drug antibodies to talquetamab will be assessed.
Number of Participants With Anti-Drug Antibodies to Teclistamab | Up to 52 Weeks
  Number of Participants with anti-drug antibodies to teclistamab will be assessed.
Overall Response Rate (ORR) | Up to 48 Weeks
  ORR is defined as the percentage of participants who have a partial response (PR) or better according to the International Myeloma Working Group (IMWG) criteria.
Clinical Benefit Rate | Up to 48 Weeks
  Clinical benefit rate (ORR + minimal response [MR]) is defined as the of participants who have a MR or better according to the IMWG criteria.
Duration of Response (DOR) | Up to 48 Weeks
  DOR is defined as the time from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria.
Time to Response | Up to 48 Weeks
  Time to response is defined as the time between date of first dose of study drug and the first efficacy evaluation that the participant has met all criteria for PR or better.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (24):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - University of California San Francisco, San Francisco, California
  - The Blavatnik Family Chelsea Medical Center at Mount Sinai, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - University Health Network UHN Princess Margaret Cancer Centre, Toronto, Ontario
- Germany (4):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Wurzburg, Würzburg
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - LUMC, Leiden
- Spain (6):
  - Hosp Clinic de Barcelona, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Germans Trias I Pujol, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Chari A, van de Donk NWCJ, Dholaria B, Weisel K, Mateos MV, Goldschmidt H, Martin TG, Morillo D, Reece D, Rodriguez-Otero P, Bhutani M, D'Souza A, Oriol A, Rosinol L, Bahlis NJ, Vishwamitra D, Skerget S, Verona RI, Bakshi K, Kang L, Prior TJ, Vandenberk L, Tolbert J, Lee S, Smit MD, Wasch R. Talquetamab plus daratumumab for the treatment of relapsed or refractory multiple myeloma in the TRIMM-2 study. Blood. 2025 Dec 11;146(24):2902-2913. doi: 10.1182/blood.2025029360. PMID 40983036
- [Derived] Pillarisetti K, Powers G, Luistro L, Babich A, Baldwin E, Li Y, Zhang X, Mendonca M, Majewski N, Nanjunda R, Chin D, Packman K, Elsayed Y, Attar R, Gaudet F. Teclistamab is an active T cell-redirecting bispecific antibody against B-cell maturation antigen for multiple myeloma. Blood Adv. 2020 Sep 22;4(18):4538-4549. doi: 10.1182/bloodadvances.2020002393. PMID 32956453